CLINICAL TRIAL: NCT01564823
Title: Adalimumab on Preventing Postoperative Recurrence of Crohn's Disease
Brief Title: Adalimumab on Preventing Post-chirurgic Recurrence on Crohn´s Disease
Acronym: APPRECIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APPRECIA
Record Dates: First submitted 2012-01-31; First posted 2012-03-28 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Crohn´s Disease
Keywords: Crohn´s disease; Metronidazole; Azathioprine; Adalimumab; post-chirurgic recurrence
MeSH Terms: conditions — Crohn Disease | interventions — Metronidazole; Azathioprine; Adalimumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole + Azathioprine. (Experimental): Metronidazole, oral intake. 250 mg/8h. 3 months. Azathioprine, 2.5 mg/weight kg/day, oral intake. All study.
  Interventions: Drug: Metronidazole; Drug: Azathioprine
- Metronidazole + Adalimumab (Active Comparator): Metronidazole Oral Intake. 250 mg/8h. During 3 months. Adalimumab Subcutaneous 160 mg and 80 mg 2wk. Then 40 mg during 2wk as maintenance.
  Interventions: Drug: Metronidazole; Drug: Adalimumab

INTERVENTIONS:
Drug: Metronidazole — Metronidazole: 250 mg/8h. 3 months.
  Other Names: Flagyl (Metronidazole)
  Arms: Metronidazole + Azathioprine.
Drug: Metronidazole — Metronidazole 250 mg/8h 3 months
  Other Names: Flagyl (Metronidazole)
  Arms: Metronidazole + Adalimumab
Drug: Azathioprine — Azathioprine: 2.5 mg/kg of weight/day. 3 months.
  Other Names: Imurel (Azathioprine)
  Arms: Metronidazole + Azathioprine.
Drug: Adalimumab — Adalimumab 160 mg then 80 mg. After 2 wk: 40 mg as maintenance.
  Other Names: Humira (Adalimumab)
  Arms: Metronidazole + Adalimumab

SUMMARY:
The present study objective is evaluate Adalimumab efficacy versus Azathioprine efficacy on prevention of endoscopic recurrence (Rutgeerts Index= 2b, 3 or 4) in Crohn´s Disease patients after 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at the time of signing informed consent.
* Patients with Crohn's disease who have undergone an ileocecal/ileocolic resection (L1 or L3). The study and the treatment must be initiated within the two first weeks after the resection (+/- 5 days).
* Patients with surgical reconstruction by ileocolic anastomosis.
* Women of childbearing age must not be breastfeeding and must have a negative urine pregnancy test and must agree to use contraceptive methods with a <1% failure rate (e.g., sexual abstinence, oral contraceptives, double barrier methods, intrauterine devices), unless they only have one partner who is sterile.
* Patients who have signed and dated the informed consent form before performing any specific screening study procedure.

Exclusion Criteria:

* Resection that requieres Temporal ileostomy.
* Urgency resection which doesn´t permit the initial assessment protocol completion.
* Resection due to inactive short indolent stenosis (<10 cm).
* Resection with mucosal macroscopic residual disease in anastomosis.
* Previous intolerance or adverse reaction (moderate or severe) to adalimumab or azathioprine.
* Any contraindications or unwillingness to perform the scheduled colonoscopies or resonances.
* Contraindications to Adalimumab treatment, among which the following are included: active tuberculosis, severe infections such as sepsis or opportunistic infections, moderate or severe heart failure (NYHA class III or IV), central nervous system demyelinating diseases, history of malignant neoplasm or autoimmune diseases.
* Severe associated Extraintestinal manifestations.
* Previous postoperative recurrence prevention treatments with adalimumab, asathiprine o mercaptopurine which resulted in failure.
* Any other disease or patient condition that according to investigator criteria, inadequates patient´s participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of endoscopic recurrences | 52 weeks after the begin of the study
  Evaluation of the effectiveness on prevention of endoscopic recurrence evaluated as changes in the Rutgeerts Index.

SECONDARY OUTCOMES:
Number of Crohns´disease remission | 24 weeks
  % of patients showing clinical remission after 24 and 52 weeks of adalimumab vs azathioprin treatment
Number of postsurgical recurrences | 52 week
  Evaluation of the Adalimumab efficiency on preventing postsurgical recurrence with Magnetic Resonance Enterography
number of hospitalized patients | 52 weeks
  Comparing hospitalization percentage in patients using adalimumab or azathioprin after 52 weeks of treatment
Concentration of activity markers | 24 weeks
  Evaluating changes in markers such as reactive c-protein, variable surface glycoprotein , faecal calprotectin, etc.
Number of surgeries | Until 52 week
  Comparing % of patients who needs surgery on Adalimumab vs Azatioprine
SIBDQ and EuroQOL indexes | 24 Weeks
  Quality of life
Number of Adverse event reports | 52 weeks
  Comparison of safety of Adalimumab versus Azatioprine.
Number of Crohns´disease remission | 52 weeks
  % of patients showing clinical remission after 24 and 52 weeks of adalimumab vs azatioprine treatment
Concentration of activity markers | 52 weeks
  Evaluating changes in markers such as reactive c-protein, VSG, faecal calprotectine, etc
SIBDQ and EuroQOL indexes | 52 weeks
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Nos, MD, Principal Investigator — Hospital Universitari i Politecnic La Fe (Valencia, Spain)
Locations (22):
- Spain (22):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Bellvitge, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital Mutua de Terrasa, Terrassa, Barcelona
  - Hospital General Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Puerto Real, Puerto Real, Cádiz
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Arquitecto Marcide, Ferrol, La Coruña
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Virgen de la Macarena, Seville, Sevilla
  - Hospital de Manises, Manises, Valencia
  - Hospital Universitari i Policlinic La Fe, Valencia, Valencia
  - Hospital Clínico, Valencia, Valencia
  - Hospital Río Hortega, Valladolid, Valladolid

REFERENCES:
- [Derived] Lopez-Sanroman A, Vera-Mendoza I, Domenech E, Taxonera C, Vega Ruiz V, Marin-Jimenez I, Guardiola J, Castro L, Esteve M, Iglesias E, Ceballos D, Martinez-Montiel P, Gisbert JP, Minguez M, Echarri A, Calvet X, Barrio J, Hinojosa J, Martin-Arranz MD, Marquez-Mosquera L, Bermejo F, Rimola J, Pons V, Nos P; Spanish GETECCU group [APPRECIA study]. Adalimumab vs Azathioprine in the Prevention of Postoperative Crohn's Disease Recurrence. A GETECCU Randomised Trial. J Crohns Colitis. 2017 Oct 27;11(11):1293-1301. doi: 10.1093/ecco-jcc/jjx051. PMID 28402454